CLINICAL TRIAL: NCT03146052
Title: Comparison Between Asymmetric (Low Dose In The Morning) And Standard Split-Dose Regimen Of Polyethylene Glycol Plus Bisacodyl For Bowel Preparation For Screening And Surveillance Colonoscopy: A Randomized Non-Inferiority Clinical Trial.
Brief Title: Comparison Between Asymmetric And Standard Split-Dose Regimen For Bowel Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Rhodense (Other)
Responsible Party: Principal Investigator, gianpiero manes, Head of the Gastroenterology Unit, ASST Rhodense
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 165-032017
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Polyps; Colon Preparation
Keywords: Colon cleansing
MeSH Terms: conditions — Polyps | interventions — Citrates; Simethicone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded endoscopists performed endoscopic procedure and evaluated colon cleansing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Asymmetric split dose preparation (Experimental): 75% of the dose is given on the day before of the procedure and 25% of the dose is given on the day of the procedure
  Interventions: Drug: PEG-4000 added with citrates and simethicone (PEG-CS) plus Bisacodyl
- Symmetric split dose preparation (Active Comparator): 50% of the dose is given on the day before of the procedure and 50% of the dose is given on the day of the procedure
  Interventions: Drug: PEG-4000 added with citrates and simethicone (PEG-CS) plus Bisacodyl

INTERVENTIONS:
Drug: PEG-4000 added with citrates and simethicone (PEG-CS) plus Bisacodyl — PEG-4000 added with citrates and simethicone (PEG-CS) (Kit contains 4 pouches, each containing 64.5gr of PEG) and bisacodyl 5 mg tablets

SUMMARY:
We aimed to compare the efficacy for bowel cleansing of a split-dose regimen with a low morning dose of PEG solution (Asymmetric; 25% of the dose is given on the day of the procedure and 75% of the dose is given on the day before) with the standard split-dose regimen in patients undergoing screening and surveillance colonoscopy using a low volume bowel preparation (2L PEG-citrate-simethicone plus Bisacodyl). We enrolled consecutive outpatients undergoing screening and surveillance colonoscopy in a randomized, single-blind, non-inferiority clinical trial. Patients were randomly assigned to: group A, asymmetric split dose regimen (1,5 L of PEG + bisacodyl the day before and 0,5 L 4 hours before colonoscopy); group B, symmetric split dose regimen (1 L of PEG + bisacodyl the day before and 1 L 5 hours before colonoscopy). Primary endpoint was the proportion of adequate bowel cleansing. Moreover, all patients filled in a nurse-administered questionnaire assessing compliance, tolerability and safety of bowel preparation.

DETAILED DESCRIPTION:
Prospective, randomized, single-blind, non-inferiority trial in adult patients undergoing screening or surveillance colonoscopy. Eligible participants were randomly assigned, according to a computer-generated list with an allocation ratio of 1:1, to receive either asymmetric or symmetric split-dose regimen of a low-volume preparation by investigators who were not involved in the enrolment process. Detailed written instructions were administered to all patients who accepted to participate. A low-fiber diet was prescribed three day before colonoscopy; participants in both groups were instructed to have a light lunch on the day before the colonoscopy and only clear liquid were allowed on the day of the exam. All endoscopic procedures were scheduled between 9:00 AM and 1:00 PM.

The preparation used in the study is a combination of a 2 L sulphate-free iso-osmotic formulation of of PEG-4000 added with citrates and simethicone (PEG-CS) (Lovol-esse; AlfaWassermann, Bologna, Italy. Kit contains 4 pouches, each containing 64.5gr of PEG, to be dissolved in 2 L of water.), and bisacodyl 5 mg tablets (Lovodyl; Alfa-Wassermann, Bologna, Italy).

All subjects were instructed to take 4 bisacodyl tablets at 4:00 PM on the day before the procedure. Subjects allocated to the asymmetric split-dose regimen group were invited to consume at 6:00 PM on the evening before the colonoscopy 3 sachets of PEG-CS in 1,5 L of water in a range from 90 to 120 minutes (about 250 mL every 15 min) and 4 hours before the scheduled procedure 1 sachets in 0,5 L of water in a range from 15 to 30 minutes. Subjects allocated to the symmetric split-dose regimen group were invited to consume at 6:00 PM on the evening before the colonoscopy 2 sachets of PEG-CS in 1 L of water in a range from 60 to 90 minutes and 5 hours before the scheduled procedure 2 sachets in 1 L of water in a range from 60 to 90 minutes.

Unblinded investigators collected demographic and clinical data with medical history. All patients filled in a nurse-administered questionnaire to assess compliance, tolerability and safety of bowel preparation.

Blinded experencied endoscopists performed endoscopic procedure in accordance with colonoscopy quality practice. Data on bowel cleansing (evaluated by using Boston Bowel Preparation Scale), endoscopic procedures and findings (i.e. cancer, polyps, diverticula) were collected.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled as outpatient for screening or surveillance colonoscopy

Exclusion Criteria:

* Inpatients
* refusal of split dose regimen for bowel preparation
* previous history of colorectal resection
* severe cardiac disease
* advanced (stage IV and V) chronic kidney disease
* pregnancy; ileus
* suspected bowel obstruction or toxic megacolon
* known inflammatory bowel disease
* known or suspected allergy to PEG.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Quality of bowel prepreparation | 2 days
  Quality of bowel prepreparation/cleanliness scored using the Boston Bowel Preparation Scale. Each segment of the colon received a score from 0 to 3, and these segment scores were summed for a total BBPS score ranging from 0 to 9. The preparation was considered adequate when BBPS score was ≥ 6 with a score with at least 2 points in any segment

SECONDARY OUTCOMES:
Adenoma detection rate | 2 days
  rate of patients with at least one adenoma
Rate of the occurrence of adverse events | 2 days
  Rate of the occurrence of adverse events (bad taste in mouth, gastric fullness, nausea or vomiting, bloating, abdominal pain, headache)
Compliance | 2 days
  Compliance was assessed by the amount of intake of study agents using a 3-point scale: 1 (100% intake), 2 (≥ 75% intake), and 3 (< 75% intake).
Tolerability | 2 days
  Tolerability was evaluated assessing how patient finds tolerable the bowel preparation by using a 4-point scale: 1 (Easy), 2 (Acceptable), 3 (Somewhat difficult), 4 (Very difficult).

CONTACTS AND LOCATIONS:
Overall Officials: Gianpiero Manes, Principal Investigator — ASST Rhodense, Garbagnate Milanese, Lombardia, Italy, 20020
Locations (1):
- ASST Rhodense, Garbagnate Milanese, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andreozzi P, De Nucci G, Bezzio C, Arena I, Devani M, Mandelli E, Morganti D, Omazzi B, Reati R, Redaelli D, Saibeni S, Manes G. Comparison of asymmetric (low morning-dose) and standard split-dose regimen of PEG plus bisacodyl for bowel preparation: A randomized controlled trial. Dig Liver Dis. 2019 Jun;51(6):837-842. doi: 10.1016/j.dld.2018.12.012. Epub 2018 Dec 28. PMID 30658942